CLINICAL TRIAL: NCT07087262
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic of SNH-119014 in Healthy Adult Volunteers
Brief Title: A Phase I Study of SNH-119014 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ScinnoHub Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SNH-119014-101
Record Dates: First submitted 2025-07-16; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Hemoglobinopathy
MeSH Terms: conditions — Hemoglobinopathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNH-119014 (Experimental)
  Interventions: Drug: SNH-119014
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SNH-119014 — study drug
  Arms: SNH-119014
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
SNH-119014 is an oral small-molecule agonist of pyruvate kinase red blood cell isozyme (PKR) being developed for the treatment of hemolytic anemias. This initial study will characterize the safety, tolerability and the pharmacokinetics/pharmacodynamics (PK/PD) of a single ascending dose and multiple ascending doses of SNH-119014 in the context of Phase 1 studies in healthy volunteers. The effects of food on the absorption of SNH-119014 will also be evaluated in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects;
* 18-45 years of age, inclusive;
* Male subjects with body weight ≥50 kg, female subjects with body weight ≥45 kg; BMI ≥18.5 and ≤28.0 kg/m2.
* Must provide written informed consent.

Exclusion Criteria:

* History of or current clinically significant circulatory system, endocrine system, nervous system, digestive system, respiratory system, urinary system, ophthalmology, hematology, immunology, psychiatry disorder, as judged by the investigator；
* Subjects who have undergone major surgery 6 months prior to screening or who plan to undergo surgery during the study period;
* Clinically significant abnormal physical examination, vital signs, chest X-ray, laboratory tests during the screening period as judged by the investigator;
* Subjects with QTcF>450 ms, or with other ECG clinically significant abnormalities during the screening period as judged by the investigator;
* Subject has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVAb), treponema pallidum antibody, or human immunodeficiency virus (HIV) antibody at screening;
* Subjects who have a known chronic liver disease, or who have clinically significant abnormal liver function test results during the screening period;
* History of urinary system diseases.
* History of dysphagia or any gastrointestinal disorder affecting drug absorption.
* History of malignancy.
* History of severe allergies or allergic to the study drug or any of its components. Serious adverse reaction or hypersensitivity to any drug or the formulation excipients.
* Failure to follow a consistent diet.
* Over 5 cups (200 ml per cup) of tea, coffee, or caffeinated beverages were consumed daily during the 3 months prior to screening.
* Consumption of a specific diet (e.g. grapefruit and grapefruit-containing products, chocolate, any food containing caffeine), or vigorous exercise, or other factors affecting drug absorption, distribution, metabolism, excretion within 48 hours before the dose of study drug.
* Subjects who have taken any drugs that alter the activity of liver enzymes and/or transporters within 28 days prior to screening.
* Females who are pregnant or lactating and subjects who are unable to use one or more nonpharmacological contraceptives.
* Subjects who have taken any prescribed or over-the-counter drug or herbal remedies or nutraceutical product within 14 days before the dose of study drug.
* Subjects who smoked more than 5 cigarettes per day during the 3 months prior to screening, or who cannot accept a smoking ban throughout the study.
* Alcohol intake >14 units per week within 6 months prior to screening (1 unit is equal to 14g of alcohol such as 360mL of beer, 45mL of 40% spirit, 150mL of wine, or a confirmed positive alcohol breath test, or alcohol prohibition is not acceptable throughout the study.
* History of drug abuse in the past 1 year prior to screening, or a confirmed positive drugs of abuse test result before randomization.
* Subjects who plan to conceive or donate sperm or eggs during the study or within 3 months after completion of study.
* Subjects has received study drug in another clinical study within 3 months before the dose of study drug.
* Subjects who have donated blood or loss ≥400 mL of blood within 3 months before the dose of study drug, or who plan to donate blood or blood components during the study or within 3 months after completion of study.
* Subjects who have received a live attenuated vaccine within 28 days before the dose of study drug.
* Subjects who cannot tolerate venipuncture, or those with a history of needle fainting or blood fainting.
* In the opinion of the investigator, the subject is not suitable for entry into the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values, Clinically Significant Physical Examination Findings, vital signs, electrocardiogram (ECG) and/or Adverse Events/Serious Adverse Events That Are Related to Treatment | up to 7 days or 20 days
  Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No